CLINICAL TRIAL: NCT02702596
Title: METRIC: Measurement, Education and Tracking in Integrated Care: Strategies to Increase Patient Engagement and Reduce Mental Health Disparities Among Hispanics
Brief Title: METRIC: Measurement, Education and Tracking in Integrated Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); University of Texas Southwestern Medical Center (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R15MD010220-01 (NIH); R15MD010220 (NIH)
Record Dates: First submitted 2016-03-03; First posted 2016-03-08 (Estimated); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBIC + DEF (Experimental): Measurement-Based Integrated Care with Depression Education Fotonovela
  Interventions: Other: Measurement-Based Integrated Care; Behavioral: Depression Education Fotonovela
- MBIC + SE (Experimental): Measurement-Based Integrated Care + Standard Education
  Interventions: Other: Measurement-Based Integrated Care; Behavioral: Standard Education

INTERVENTIONS:
Other: Measurement-Based Integrated Care — Measurement-Based Integrated Care (MBIC) synthesizes the science of integrated health care and incorporates the strategies of measurement-based care. concept of MBIC for the treatment of depression includes: systematic assessment of symptoms, antidepressant treatment side effects and medication adherence and incorporation of a Depression Care Manager (DCM) to track patients and keep them engaged in care using behavioral interventions
Behavioral: Depression Education Fotonovela — Depression education that uses a unique, culturally adapted depression fotonovela titled "Secret Feelings" developed by Cabassa, Molina and Baron (2012). The fotonovela is a popular comic-book style pamphlet that portrays a dramatic story using photographs and dialogue bubbles, which has become an effective tool for engaging Hispanic audiences and increasing knowledge about specific health issues
  Arms: MBIC + DEF
Behavioral: Standard Education — The the use of a pamphlet to educate people about depression.
  Arms: MBIC + SE

SUMMARY:
The proposed study seeks to establish the feasibility of universal screening for depression in an adult primary care safety net setting, measure the effectiveness of a culturally appropriate depression education intervention to reduce stigma and increase uptake in depression treatment among Hispanics, and implement a Measurement-Based Integrated Care (MBIC) model with collaborative, multi-disciplinary treatment and culturally tailored care management strategies.

DETAILED DESCRIPTION:
Specific Aim 1: Examine the specific effects of a Depression Education Fotonovela (DEF) to increase knowledge of depression, reduce stigma and increase engagement in depression treatment among Hispanic patients.

Specific Aim 2: Evaluate the impact of Measurement-Based Integrated Care (MBIC) for the treatment of depression in one community-based Federally Qualified Health Centers (FQHC) in North Texas whose patient population is majority Hispanic.

Specific Aim 3: Examine the feasibility of universal screening and accurate detection of depression among adult primary care patients utilizing innovative iPad Depression Screening technology.

ELIGIBILITY:
Inclusion Criteria:

* Adult primary care patients
* Hispanic
* Meets diagnostic criteria for depression

Exclusion Criteria:

* currently in treatment for depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who engage in depression treatment | baseline to one month post education session
Change in PHQ-9 (depressive symptoms) scores | baseline compared to one year post enrollment

SECONDARY OUTCOMES:
Number of primary care patients screened for depression using the iPad technology | two year participant enrollment period

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Sanchez, PhD, Principal Investigator — University of Texas at Arlington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sanchez K, Eghaneyan BH, Killian MO, Cabassa LJ, Trivedi MH. Depression education fotonovela for engagement of Hispanic patients in treatment: a randomized clinical trial. BMC Psychiatry. 2021 Dec 23;21(1):635. doi: 10.1186/s12888-021-03641-0. PMID 34949169
- [Derived] Sanchez K, Eghaneyan BH, Killian MO, Cabassa L, Trivedi MH. Measurement, Education and Tracking in Integrated Care (METRIC): use of a culturally adapted education tool versus standard education to increase engagement in depression treatment among Hispanic patients: study protocol for a randomized control trial. Trials. 2017 Aug 3;18(1):363. doi: 10.1186/s13063-017-2109-y. PMID 28774339